CLINICAL TRIAL: NCT05047146
Title: The Clinicopathological and Prognostic Factors of Hepatocellular Carcinoma; 10 Years' Tertiary Center Experience in Egypt
Status: Completed | Type: Observational
Sponsor: Sadat City University (Other)
Responsible Party: Principal Investigator, Mahmoud Samy Abdallah, Lecturer of Clinical Pharmacy, Sadat City University
Other Study IDs: 00246/2021
Record Dates: First submitted 2021-09-02; First posted 2021-09-16 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Morphological classifications of HCC — Morphological classifications of Hepatocellular carcinoma

SUMMARY:
This study aimed at study the clinical and pathological criteria of Hepatocellular carcinoma to keep with new challenging in diagnosis and morpho-molecular classifications

ELIGIBILITY:
Inclusion Criteria:

* All pathologically proven Hepatocellular Carcinoma

Exclusion Criteria:

* Other malignant tumors than Hepatocellular Carcinoma
* Benign tumor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCC cases from a single tertiary center eligible for pathological analysis as a primary tool
Sampling Method: Non-Probability Sample
Enrollment: 530 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Clinicopathological factors of Hepatocellular Carcinoma | 10 years
  Serum alpha-fetoprotein (AFP) level
Clinicopathological factors of Hepatocellular Carcinoma | 10 years
  Tumor size and focality
Clinicopathological factors of Hepatocellular Carcinoma | 10 years
  Vascular invasion
Clinicopathological factors of Hepatocellular Carcinoma | 10 years
  Pathologic stage and grade
Clinicopathological factors of Hepatocellular Carcinoma | 10 years
  The reserve of background liver

CONTACTS AND LOCATIONS:
Locations (1):
- National Liver Intitute, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
sharing will be by website or google after paper publication
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Sweed D, Sweed E, Moaz I, Mosbeh A, Fayed Y, Elhamed SMA, Sweed E, Macshut M, Abdelsattar S, Kilany S, Saied SA, Badr R, Abdallah MS, Ehsan N. The clinicopathological and prognostic factors of hepatocellular carcinoma: a 10-year tertiary center experience in Egypt. World J Surg Oncol. 2022 Sep 19;20(1):298. doi: 10.1186/s12957-022-02764-2. PMID 36117166